CLINICAL TRIAL: NCT04979247
Title: Intravenous Oliceridine and Opioid-related Complications: VOLITION: A Multicenter Pilot Cohort Study
Brief Title: Intravenous Oliceridine and Opioid-related Complications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-684
Record Dates: First submitted 2021-07-16; First posted 2021-07-28 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Major Surgery
MeSH Terms: interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oliceridine (Experimental): Patients receive Oliceridine for pain control.
  Interventions: Drug: Oliceridine

INTERVENTIONS:
Drug: Oliceridine — Near the end of surgery, patients will be given ≤1.5 mg of oliceridine as a bolus. Postoperatively, patient-controlled analgesia (PCA) will be started with no background infusion, demand doses of 0.35 mg, with a 6 minute lock-out. Additional boluses (≤1 mg) of oliceridine will be given as deemed necessary (based on NRS score and clinical assessment of the patient) as soon as 15 minutes after the initial 1.5 mg loading dose. In addition to supplemental 1 mg bolus doses, the PCA demand dose can be increased to a maximum of 0.5 mg oliceridine.

SUMMARY:
The investigator will evaluate the side effects of oliceridine.

DETAILED DESCRIPTION:
The investigator will evaluate the side effects of oliceridine. Limited information suggests that oliceridine may cause fewer side effects than the standard opioids given post surgery. Oliceridine is effective for treating acute pain, and is approved by the FDA. Patients will wear a device that continuously monitors breathing. Data from this monitor will be blinded to the clinical staff. Primary Aims include: The investigators will evaluate the proportion of patients having an adjudicated meaningful respiratory compromise with a specified precision of 0.15 using a 95% confidence interval at 24 hours post first study dose.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* American Society of Anesthesiologists physical status 1-4
* Scheduled for major noncardiac surgery expected to last at least 2 hours
* Expected to remain hospitalized at least two postoperative nights
* Scheduled for general endotracheal, spinal anesthesia, or the combination
* Expected to require substantial opioid analgesia, defined as ≥20 mg morphine equivalents
* Expected to have patient-controlled intravenous analgesia.

Exclusion Criteria:

* Are demented or otherwise cannot provide valid consent
* Have contraindications to oliceridine
* Used legal or illegal opioids chronically, defined as >15 mg morphine equivalents for >15 days during the month before consenting by history
* Have language, vision, or hearing impairments that may compromise continuous ventilation monitoring
* Have planned epidural anesthesia/analgesia
* Planned spinal morphine administration
* Are designated Do Not Resuscitate, hospice, or receiving end of life therapy
* Are expected to require postoperative mechanical ventilation or ICU admission
* Are expected to receive intrathecal opioids
* Are expected to receive gabapentin, pregabalin or other analgesic adjuvants
* Use oxygen at home
* Are unwilling or unable to comply fully with study procedures (including not tolerating the capnography cannula)
* Are known to be pregnant or breastfeeding
* Use CPAP at home
* Have previously participated in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Number of patients who have respiratory compromise. | 24 hours post first study dose.
  Respiratory compromise will be defined by a collapsed (one or more) composite of 1) end-tidal carbon dioxide <15mmHg for ≥3 minutes; 2) respiratory rate ≤5 breaths/minute for ≥3 minutes; 3) SpO2 ≤ 85% for ≥3 minutes; 4) Apnea episode lasting >30 seconds; 5)any serious respiratory event.

SECONDARY OUTCOMES:
Cumulative duration of oxygen saturation < 90% | 48 hours post first study dose.
  The sum of minutes with SpO2<90% from monitoring data
Cumulative duration of respiratory rate < 8 breaths/ minute | 48 hours post first study dose.
  The sum of minutes with respiratory rate < 8 from monitoring data

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Principal Investigator — The Cleveland Clinic
Locations (3):
- United States (3):
  - Wake Forest Bapist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio

REFERENCES:
- [Derived] Sessler DI, Ayad S, Bakal O, Disher NS, Duran JA, Weingarten TN, Dahan A, Demitrack MA, Kim J, Khanna AK; VOLITION Study Team. Oliceridine for postoperative pain and opioid-related complications: The intravenous oliceridine and opioid-related complications (VOLITION) prospective cohort study. J Clin Anesth. 2025 Jul;105:111870. doi: 10.1016/j.jclinane.2025.111870. Epub 2025 May 29. PMID 40446423